CLINICAL TRIAL: NCT02322827
Title: Adherence & Health Outcome Differences Amongst HIV Infected Patients Prescribed a Single Tablet Regimen (STR) Versus Multi Tablet Regimen (MTR).
Brief Title: Adherence & Health Outcome Differences Amongst HIV Infected Patients Prescribed HAART
Acronym: HOST
Status: Completed | Type: Observational
Sponsor: Olayemi Osiyemi MD (Other)
Responsible Party: Sponsor-Investigator, Olayemi Osiyemi MD, President, Triple O Research Institute PA
Organization: Triple O Research Institute PA (Other)
Other Study IDs: IN-US-236-1642
Record Dates: First submitted 2014-11-25; First posted 2014-12-23 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Acquired Immunodeficiency Syndrome; Human Immunodeficiency Virus Type
Keywords: hiv/aids
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- single tablet regimen: Subjects whose most recent antiretroviral therapy consist of a single tablet regimen
- multiple tablet regimen: Subjects whose most recent antiretroviral therapy consist of multi tablet regimen

SUMMARY:
This study is designed to see how HIV infected patients perform when taking a single fixed dose HIV medication compared to a regimen with multiple tablets. The study is also going to be looking at the differences in complications between the two groups.

DETAILED DESCRIPTION:
This is a phase IV retrospective chart review of HIV infected patients in a private Infectious disease practice in West Palm Beach, FL. This chart review will assign patients into one of two groups based on their antiretroviral regimen: single tablet regimen (STR) versus multi tablet regimen (MTR). Up to 650 patient charts will be reviewed but only about 500 patients are needed for statistical analysis.

The primary objective is to look at the proportion of patients with an adherence rate greater than or equal to 95% in subjects prescribed STR versus a MTR.

Secondary Objectives:

* Differences in emergency room visits, hospitalization and readmission in patients taking a STR vs. a MTR
* Proportion of patients with HIV viral load less than 50copies/microliter
* Incidence of new onset or worsening hyperlipidemia in patients taking a STR versus a MTR
* Incidence of acute renal insufficiency
* Compare the absolute CD4 number increase between a STR and a MTR
* Compare monthly copay amounts in patients taking a STR versus a MTR
* Identify the incidence of opportunistic infections in patients taking a STR versus a MTR

ELIGIBILITY:
Inclusion Criteria:

* Male or Female (gender at birth), age 18 years or older
* Documented HIV-1 infection by western blot or HIV viral load
* Prescribed antiretroviral therapy, either STR (single tablet regime) or MTR (multi tablet regimen) for at least 6 months
* Patients should have a minimum of 3 office visits

Exclusion Criteria:

* Patients who were evaluated in the hospital but never came to the clinic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are HIV infected and taking antiretroviral therapy
Sampling Method: Non-Probability Sample
Enrollment: 445 (Actual)
Dates: Start 2014-11; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Compare the proportion of patients with an adherence rate greater than or equal to 95% in subjects taking a STR versus a MTR | 1 year

SECONDARY OUTCOMES:
compare differences in ER visits, hospitalizations and readmissions in patients taking a STR versus a MTR | 2 years
  composite
Compare proportion of subjects with viral load less than 50 copies/microL | 1year
Identify the incidence of new onset or worsening hyperlipidemia in subjects taking a TR versus a MTR | 2 years
Identify the incidence of acute renal insufficiency in subjects taking a STR versus a MTR | 2 years
Compare the absolute CD4 number increase between a STR and a MTR | 1 year
Compare monthly copay amounts in patients prescribed STR and MTR | 1 year
Identify the incidence of opportunistic infections in subjects taking a STR versus a MTR | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Olayemi Osiyemi, M.D., Principal Investigator — Triple O Research Institute PA
Locations (1):
- Triple O Research Institute PA, West Palm Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided